CLINICAL TRIAL: NCT05660720
Title: A Randomized, Blinded, Placebo- and Positive-Controlled, Four-Period, Crossover-Design Thorough QT/QTc (TQT) Study to Evaluate the Effect of Orelabrutinib on Cardiac Repolarization in Healthy Subjects
Brief Title: Evaluate the Effect of Orelabrutinib on Cardiac Repolarization in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00120
Record Dates: First submitted 2022-11-11; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Healthy Subject
MeSH Terms: interventions — orelabrutinib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Orelabrutinib tablet 150 mg (study drug) and placebo 250 mg (orelabrutinib tablet simulator) (Experimental): The subjects will be dosed once on Day1 or Day6 or Day11 or Day16 according to randomization.
  Interventions: Drug: Orelabrutinib and placebo (orelabrutinib tablet simulator)
- Orelabrutinib 400 mg (study drug) (Experimental): The subjects will be dosed once on Day1 or Day6 or Day11 or Day16 according to randomization.
  Interventions: Drug: Orelabrutinib
- Placebo 400mg (orelabrutinib tablet simulator) (Placebo Comparator): The subjects will be dosed once on Day1 or Day6 or Day11 or Day16according to randomization.
  Interventions: Drug: Placebo (orelabrutinib tablet simulator)
- Moxifloxacin hydrochloride 400 mg (Active Comparator): he subjects will be dosed once on Day1 or Day6 or Day11 or Day16 according to randomization.
  Interventions: Drug: Moxifloxacin hydrochloride

INTERVENTIONS:
Drug: Orelabrutinib and placebo (orelabrutinib tablet simulator) — Orelabrutinib will be administered as 3 tablets (150mg) and placebo as 5 tablets (250mg)
  Arms: Orelabrutinib tablet 150 mg (study drug) and placebo 250 mg (orelabrutinib tablet simulator)
Drug: Orelabrutinib — Orelabrutinib will be administered as 8 tablets (400mg)
  Arms: Orelabrutinib 400 mg (study drug)
Drug: Placebo (orelabrutinib tablet simulator) — Placebo will be administered as 8 tablets (400mg).
  Arms: Placebo 400mg (orelabrutinib tablet simulator)
Drug: Moxifloxacin hydrochloride — Moxifloxacin hydrochloride will be administered as 1 tablet (400mg)
  Arms: Moxifloxacin hydrochloride 400 mg

SUMMARY:
This is A Randomized, Blinded, Placebo- and Positive-Controlled, Four-Period, Crossover-Design Thorough QT/QTc (TQT) Study to Evaluate the Effect of Orelabrutinib on Cardiac Repolarization in Healthy Subjects

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo- and positive-controlled, four-period, crossover clinical study. A double-blind design is used for administration of orelabrutinib tablet and placebo, and an open-label design is used for moxifloxacin hydrochloride tablet.Subjects who meet all inclusion criteria and do not meet any of the exclusion criteria are randomly assigned to one of 12 treatment sequences, and each treatment sequence includes 4 periods, with a 5-day washout period between treatment periods. The subject will complete all the visit examinations on Day 17 after the first dose, then will be discharged from the study site, and will receive telephone follow-up on Day 8 ± 2 after the last dose date. If a subject has clinically significant abnormal examination results when discharging from the study site after the last dose, on-site follow-up is essential to track the abnormal examination results, or otherwise, only telephone follow-up is required.

ELIGIBILITY:
Inclusion Criteria

1. After being informed and understanding of the trial process and possible adverse reactions of the drug, the subjects voluntarily signed an informed consent form (ICF) and confirmed their participation in all study procedures;
2. Healthy subjects aged 18-45 years (inclusive) at the time of signing the informed consent;
3. Weight of subjects ≥50.0 kg and ≤100.0 kg; Body mass index (BMI) ≥19.0 kg/m2 and ≤ 30.0 kg/m2, BMI= weight (kg)/height 2 (m2);
4. Subjects do not have clinically meaningful medical history and various examinations including physical examination, vital signs, laboratory tests or ECG, and the results are normal or abnormal without clinical significance judged by investigators.
5. Eligible fertile subjects (male and female) must agree to abstain from sex (avoid heterosexual sex) or use effective contraceptives with an annual contraceptive failure rate of less than 1% during the trial period until 3 months after the end of the trial.

Exclusion Criteria

1. History of any clinically serious disease like heart, liver, kidney, gastrointestinal tract, blood and respiratory system, immune system etc, with a history of fainting during acupuncture or injection or when seeing blood, or cannot tolerate venipuncture;
2. Abnormal renal ,liver and pancreas function;
3. Low blood pressure (systolic blood pressure<90 mmHg; diastolic blood pressure<60 mmHg) or hypertension (systolic blood pressure ≥ 140 mmHg; diastolic blood pressure ≥ 90 mmHg);
4. Prolonged QTc interval that is at risk of causing torsade de pointes (TdP) requires drug treatment or other heart related abnormalities require drug treatment;
5. The average value of three repetitions of 12 lead ECG at screening and before the first administration exceeded the standard: PR>220 ms, QRS>120 ms, HR<50 bpm, QTcF>450 ms (male and female), and any ECG abnormality with clinical significance determined by the investigator at screening;
6. With a history of dysphagia or any gastrointestinal disease that affects drug absorption;
7. With a history of drug or food allergy, or a history of specific allergies (asthma, urticaria, eczema, etc.); or allergic to moxifloxacin or other fluoroquinolones;
8. Within 3 months before screening, those who have undergone surgery, have smoked more than 5 cigarettes or e-cigarettes daily, with a history of drug abuse or illicit drug use, or plan to undergo surgery during the study period, or with positive results of urine drug test at screening;
9. Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health products within 14 days before the first dose;
10. People with positive results of one or more of the following tests: hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), HIV antigen/antibody joint test (HIV Ab), Treponema pallidum antibody (TP Ab) and COVID-19 at screening;
11. Within 1 month before screening, those who have received anticoagulant therapy or thrombin inhibitor and/or antiplatelet therapy, any drug that inhibits or induces the metabolism of a drug by the liver;
12. Those who have frequently used alcohol within 6 months before screening, or those who are unable to abstain from alcohol during the study period, or those who have positive results of breath alcohol test at the time of screening;
13. Within 7 days before screening those who have drunk excessive tea, coffee or caffeinated beverages, or who have eaten fruits or food that affect metabolic enzymes, within 1 months before screening who are used to beverages or food rich in xanthine ingredients, and those who are unable to abstain from such beverages, fruits or food mentioned above during the whole study period;
14. Those who have participated in 4 or more clinical trials during the past one year; who have taken other study drugs or participated in other drug clinical trials within 3 months before screening;
15. Those who have donated blood or plan to donate blood within 3 months before screening, or have received blood transfusion within 4 weeks before screening;
16. Those who have been vaccinated within 4 weeks before screening, or plan to get vaccinated during the study period;
17. Women who are pregnant or breastfeeding, or have positive results of serum human chorionic gonadotropin (HCG) test before the first dose;
18. Those who disagree to discontinue strenuous exercises from the date of signing the ICF to the end of the trial (including non-hospitalization period);
19. Those who cannot complete this study due to other reasons or who have clinically significant lab abnormalities as determined by the investigator, or who are not suitable for this study as assessed by the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-19 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Placebo-corrected change-from-baseline QTcF interval | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.

SECONDARY OUTCOMES:
Change-from-baseline QTcF, PR, and QRS intervals | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.
Change-from-baseline HR | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.
Placebo-corrected change-from-baseline PR, and QRS intervals | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.
Placebo-corrected change-from-baseline HR | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.
Categorical outliers for QTcF, PR, and QRS | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.
Categorical outliers for HR | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.
Frequency of treatment-emergent changes of T-wave morphology and U-waves presence | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Extraction of Holter ECGs from 1 h pre-dose to 24 h post-dose in each period.
Tmax of Orelabrutinib after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
Cmax of Orelabrutinib after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
AUC of Orelabrutinib after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
T1/2 of Orelabrutinib after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
CL/F of Orelabrutinib after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
Vz/F of Orelabrutinib after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
Tmax of moxifloxacin after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
Cmax of moxifloxacin after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
AUC of moxifloxacin after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
T1/2 of moxifloxacin after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
CL/F of moxifloxacin after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
Vz/F of moxifloxacin after single dose | Day1, Day2, Day6, Day7, Day11, Day12, Day16 and Day17
  Plasma samples will be collected from all the subjects for PK analysis. For each period, venous blood will be collected within 30 min pre-dose, and 0.5 h, 1.0 h, 2.0 h, 3.0 h, 4.0 h, 6.0 h, 8.0 h, 12.0 h, and 24.0 h post-dose.
Serious adverse events (SAEs) occurring from administration of drugst to follow-up period or early withdrawal, incidence of treatment-emergent adverse events | Through study completion, an average of 1 year
  SAE and TEAE

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Boren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No